CLINICAL TRIAL: NCT04749095
Title: Can Bilateral Erector Spinae Plane Block Minimize Perioprative Opioid Consumption and Provide Satisfactory Analgesia for Lumbar Spine Fusion Surgery? A Randomized Controlled Study
Brief Title: Erector Spinae Plane Block Analgesia for Lumbar Spine Fusion Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Baher Said Elshahat Mohamed Abdelhady, Principal Investigator, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: erector spinae plane block
Record Dates: First submitted 2021-02-05; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector block (Active Comparator)
  Interventions: Drug: Erector spinae plane block
- sham block (Active Comparator)
  Interventions: Drug: sham subcutaneous infiltration

INTERVENTIONS:
Drug: Erector spinae plane block — bilateral ESP block will be injected with 20 ml of 0.25% bupivacaine
  Arms: Erector block
Drug: sham subcutaneous infiltration — bilateral ESP block will be injected with 20 ml of normal saline
  Arms: sham block

SUMMARY:
The purpose of this study was to investigate the effect of a bilateral ultrasound guided erector spinae plane block on the pain scores and opoid utiliziation in fusion surgery of the lumbar spine.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists class I-III adult patients
* BMI less than or equal 35 kg/m2

Exclusion Criteria:

* Patient refusal
* unable to give consent
* age < 18 or > 65
* BMI more than 35 kg/m2
* known allergy to the study medication
* coagulopathies or on anticoagulant medications
* hepatic insufficiency
* renal insufficiency
* chronic opioid use

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Analgesia | Up to 24 hours after surgery
  Numerical rating scale of pain every 6 hours